CLINICAL TRIAL: NCT01582503
Title: A Phase IIb, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, and Dosing Regimens of MEMP1972A in Adults With Allergic Asthma Who Are Inadequately Controlled on Inhaled Corticosteroids and a Second Controller (COSTA)
Brief Title: A Study of MEMP1972A in Patients With Allergic Asthma Inadequately Controlled on Inhaled Steroids And A Second Controller (COSTA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GB27980; 2011-003997-10 (EudraCT Number)
Record Dates: First submitted 2012-04-19; First posted 2012-04-20 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- MEMP1972A 150 mg (Experimental)
  Interventions: Drug: MEMP1972A
- MEMP1972A 300 mg (Experimental)
  Interventions: Drug: MEMP1972A
- MEMP1972A 450 mg (Experimental)
  Interventions: Drug: MEMP1972A
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: MEMP1972A — Subcutaneous repeating dose
  Arms: MEMP1972A 300 mg
Drug: MEMP1972A — Subcutaneous repeating dose
  Arms: MEMP1972A 450 mg
Drug: MEMP1972A — Subcutaneous repeating dose
  Arms: MEMP1972A 150 mg
Drug: placebo — Subcutaneous repeating dose
  Arms: Placebo

SUMMARY:
This randomized, double-blind, placebo-controlled study will evaluate the efficacy and safety of 3 dosing regimens of MEMP1972A in patients with allergic asthma who remain inadequately controlled on chronic therapy with high dose inhaled corticosteroids and a second controller medication.Patients will be randomized to 4 Arms to receive subcutaneous repeating dose of either MEMP1972A 150 mg, 300 mg, or 450 mg, or placebo. Patients will continue their usual asthma medication throughout the study. Anticipated time on study treatment is 36 weeks, with a 48-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18 to 75 years of age inclusive
* Body weight >/= 40 kg
* Physician's diagnosis of asthma for at least 12 months
* Evidence of documented bronchodilator reversibility as defined by protocol
* Prebronchodilator FEV1 >/= 40% and </= 80% predicted at Visit 1
* Required daily use of ICS and a second controller for a minimum of 3 consecutive months prior to Visit 1
* History of at least one protocol-defined asthma exacerbation in the 18 months prior to Visit 1
* Inadequately controlled asthma despite compliance with asthma controller therapy

Exclusion Criteria:

* Asthma exacerbation requiring systemic steroids in the 30 days prior to Visit 1
* Pre-existing active lung disease other than asthma
* Any infection
* Clinically significant medical disease that is uncontrolled despite treatment or is likely to require a change in therapy during study or is of unknown etiology
* Known immunodeficiency, including but not limited to HIV infection, regardless of treatment status
* Current substance abuse
* Former smoker with >10 pack-year history or current smoker; former smokers must have stopped smoking more than 12 months prior to Visit 1
* History of anaphylaxis
* Pregnant and lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 578 (Actual)
Dates: Start 2012-04; Primary Completion 2014-05 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Rate of protocol-defined asthma exacerbations (new or increased asthma symptoms that lead to treatment with systemic corticosteroids or to hospitalization) from baseline to Week 36 | 36 weeks

SECONDARY OUTCOMES:
Relative change in pre-bronchodilator FEV1 (volume) | from baseline to Week 12
Relative change in FEV1 (volume) | from baseline to Week 36
Change in asthma symptoms | from baseline to Week 12
Change in asthma symptoms | from baseline to Week 36
Proportion of "well-controlled" weeks (no nighttime awakenings due to asthma symptoms and </= 2 days of SABA use per weeks, as documented by patient diary) from Week 24 to Week 36 | 12 weeks
Safety: Incidence of adverse events | 48 weeks
Incidence of anti-therapeutic antibodies (ATAs) | 84 weeks
Pharmacokinetics: Area under the concentration-time curve (AUC) | Pre- and post-dose Weeks 0, 4, 12, 24 and 36

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (120):
- United States (49):
  - Birmingham, Alabama
  - Bakersfield, California
  - Costa Mesa, California
  - Fountain Valley, California
  - Long Beach, California
  - Mission Viejo, California
  - Rancho Cordova, California
  - Redwood City, California
  - Stockton, California
  - Torrance, California
  - Upland, California
  - Centennial, Colorado
  - Denver, Colorado
  - New Haven, Connecticut
  - Tampa, Florida
  - Winter Park, Florida
  - Albany, Georgia
  - Twin Falls, Idaho
  - Normal, Illinois
  - River Forest, Illinois
  - Iowa City, Iowa
  - Overland Park, Kansas
  - Louisville, Kentucky
  - Baltimore, Maryland
  - St Louis, Missouri
  - Bellevue, Nebraska
  - Omaha, Nebraska
  - Edison, New Jersey
  - Teaneck, New Jersey
  - The Bronx, New York
  - Winston-Salem, North Carolina
  - Canton, Ohio
  - Centerville, Ohio
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Medford, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Warwick, Rhode Island
  - Charleston, South Carolina
  - El Paso, Texas
  - San Antonio, Texas
  - Waco, Texas
  - Murray, Utah
  - Fairfax, Virginia
  - Spokane, Washington
  - Greenfield, Wisconsin
- Argentina (7):
  - Buenos Aires
  - Mendoza
  - Quilmes
  - Rosario
  - Salta
  - San Juan Bautista
  - San Miguel de Tucumán
- Belgium (3):
  - Gembloux
  - Halen
  - Leuven
- Bulgaria (6):
  - Pleven
  - Plovdiv
  - Rousse
  - Sofia
  - Stara Zagora
  - Varna
- Canada (4):
  - Vancouver, British Columbia
  - Mississauga, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
- Germany (10):
  - Berlin
  - Bochum
  - Coswig
  - Freiburg im Breisgau
  - Geesthacht
  - Jena
  - Landsberg
  - Magdeburg
  - Mainz
  - Münster
- Hungary (3):
  - Balassagyarmat
  - Debrecen
  - Mosonmagyaróvar
- Mexico (3):
  - Guadalajara
  - México
  - Nuevo León
- New Zealand (6):
  - Auckland
  - Aucklund
  - Christchurch
  - Dunedin
  - Hamilton
  - Wellington
- Peru (3):
  - Lima
  - Miraflores
  - Piura
- Poland (10):
  - Bialystok
  - Katowice
  - Kielce
  - Krakow
  - Lublin
  - Poznan
  - Skierniewice
  - Tarnów
  - Warsaw
  - Wroclaw
- Romania (5):
  - Brasov
  - Bucharest
  - Cluj-Napoca
  - Craiova
  - Deva
- Russia (4):
  - Moscow
  - S. Petersburg
  - Saint Petersburg
  - Smolensk
- Ukraine (7):
  - Dnipro
  - Dnipropetrovsk
  - Ivano-Frankivsk
  - Kiev
  - Kyiv
  - Lviv
  - Odesa

REFERENCES:
- [Derived] Harris JM, Maciuca R, Bradley MS, Cabanski CR, Scheerens H, Lim J, Cai F, Kishnani M, Liao XC, Samineni D, Zhu R, Cochran C, Soong W, Diaz JD, Perin P, Tsukayama M, Dimov D, Agache I, Kelsen SG. A randomized trial of the efficacy and safety of quilizumab in adults with inadequately controlled allergic asthma. Respir Res. 2016 Mar 18;17:29. doi: 10.1186/s12931-016-0347-2. PMID 26993628